CLINICAL TRIAL: NCT05437627
Title: Computerized Based Analysis for Detection and Severity Assessment of Stuttering
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Fathy, principal investigator, Assiut University
Other Study IDs: Stuttering using Computer
Record Dates: First submitted 2022-06-26; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Stuttering
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group:: Study Group: This will be consisted of sixty (60) stuttering patients. They will be divided into 2 subgroups; children group 30 patients with age ranges from (10-18y) and adult group 30 patients with age ranges from (19-30y)
  Interventions: Diagnostic Test: The Arabic version of Stuttering Severity Instrument-3 (ASSI3) for children and adults
- Control Group: Control Group: This will be consisted of sixty (60) subjects who have normal fluency. They will be selected from the relative of the patients attending to the outpatient clinic and will be matched for age, sex and socioeconomic state with the patients group.

INTERVENTIONS:
Diagnostic Test: The Arabic version of Stuttering Severity Instrument-3 (ASSI3) for children and adults — Assessment of stuttering severity: The Arabic version of Stuttering Severity Instrument-3 (ASSI3) for children and adults will be applied for assessment of severity of stuttering. (3).
  Automatic detection and severity assessment of stuttering using MATLAB version 8.1.0.604 R2013a (7). Stuttering detection system has three main steps which are acoustic processing, feature extraction and classification/recognition
  Other Names: A. Acoustic voice analysis; B. Spectral analysis:; Automatic detection and severity assessment of stuttering
  Groups: Study Group:

SUMMARY:
In the light of previous attempts to design and develop automated and objective measures for automatic speech recognition system that detects disfluent speech and assess its severity, yet fully automated measurement of stuttered speech is not available. This study was triggered by the need to design and develop a simple and reliable computerized tool for identification of stuttering and measurement for its severity. Therefore, the aim of this study is to develop a user interface that can work on windows system for the adopted stuttering recognition model which can be used in clinical practice by physicians and therapists.

DETAILED DESCRIPTION:
Stuttering is a speech disorder in which the normal flow of speech is disrupted by occurrences of dysfluencies, such as repetition, prolongations and blocks (1). Features that have been found to differ between stutterers and nonstutterers are rate of speech and frequency of dysfluent utterances (2).

An Arabic version of stuttering severity instrument (A-SSI) is used to assess the stuttering severity In it, the overall severity score of stuttering is measured by combining the scores of percentages of Stuttered Syllables (%SS), Mean Duration of the Three Longest Stuttering Events (MDTLSE), and Physical Concomitants (PC) (3).

The subjective assessment methods of stuttering are; time-consuming, prone to error, subjective (4), so it is better to automate the measurement of disfluencies using speech recognition technologies and computational intelligence (5).

Speech recognition executes a task similar to what the human brain undertakes (6). Stuttering detection system has three main steps which are acoustic processing, feature extraction and classification/recognition (7). the speech signals are pre-processed (8), and certain features are extracted from them by signal processing techniques, e.g. Mell frequency cepstral coefficients (MFCC) (9). (MFCC) is considered the most popular used feature extraction technique (10).

The classification process contains two steps; training and testing (11). In training process, data is labeled based on the classes and a model is learned. In testing phase: the model is tested and computed the accuracy, sensitivity, and specificity of the classification models (11). Finally, stuttering from non-stuttering speech will be recognized and separated (5) also to assess the severity of stuttered speech.

ELIGIBILITY:
Inclusion Criteria:

1. Age: from 10 to 30 years old.
2. Gender: both sexes will be included in the study.
3. The participants in the study group suffering from developmental stuttering (stuttering symptoms was of early childhood onset, intermittent course and dated since early childhood) seeking speech therapy
4. Have language aptitudes coping with his or her chronological age.

Exclusion Criteria:

* 1. Presence of any other speech or language disorders. 2. Mental Retardation. 3. Poor scholastic performances. 4. Presence of any psychiatric or neurologic disorders.

Ages: 10 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study will be included one hundred twenty (120) subjects; age ranges (10-30 years). They will be recruited from the outpatient clinic of Phoniatric Unit, Assiut University Hospital. The study is supposed to be conducted in one up to 2 years. They will be divided into two groups:
  1. Study Group: This will be consisted of sixty (60) stuttering patients. They will be divided into 2 subgroups; children group 30 patients with age ranges from (10-18y) and adult group 30 patients with age ranges from (19-30y)
  2. Control Group: This will be consisted of sixty (60) subjects who have normal fluency. They will be selected from the relative of the patients attending to the outpatient clinic and will be matched for age, sex and socioeconomic state with the patients group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of stuttering severity: | baseline
  using both subjective method as The Arabic version of Stuttering Severity Instrument-3 (ASSI3) for children and adults and objective method asAutomatic detection and severity assessment of stuttering

REFERENCES:
- [Background] Bakker K, Brutten GJ. Speech-related reaction times of stutterers and nonstutterers: diagnostic implications. J Speech Hear Disord. 1990 May;55(2):295-9. doi: 10.1044/jshd.5502.295. PMID 2329792
- [Background] Andrews G, Craig A, Feyer AM, Hoddinott S, Howie P, Neilson M. Stuttering: a review of research findings and theories circa 1982. J Speech Hear Disord. 1983 Aug;48(3):226-46. doi: 10.1044/jshd.4803.226. PMID 6353066
- [Background] Yairi E. Subtyping stuttering I: a review. J Fluency Disord. 2007;32(3):165-96. doi: 10.1016/j.jfludis.2007.04.001. Epub 2007 Apr 24. PMID 17825668
- [Background] Prasse JE, Kikano GE. Stuttering: an overview. Am Fam Physician. 2008 May 1;77(9):1271-6. PMID 18540491
- [Background] SHERMAN D. Clinical and experimental use of the Iowa Scale of Severity of Stuttering. J Speech Hear Disord. 1952 Sep;17(3):316-20. doi: 10.1044/jshd.1703.316. No abstract available. PMID 13053555
- [Background] O'Brian S, Packman A, Onslow M, O'Brian N. Measurement of stuttering in adults: comparison of stuttering-rate and severity-scaling methods. J Speech Lang Hear Res. 2004 Oct;47(5):1081-7. doi: 10.1044/1092-4388(2004/080). PMID 15603463
- [Background] Enderby PM, John A. Therapy outcome measures in speech and language therapy: comparing performance between different providers. Int J Lang Commun Disord. 1999 Oct-Dec;34(4):417-29. doi: 10.1080/136828299247360. PMID 10884909
- [Background] Prins D, Ingham RJ. Evidence-based treatment and stuttering--historical perspective. J Speech Lang Hear Res. 2009 Feb;52(1):254-63. doi: 10.1044/1092-4388(2008/07-0111). Epub 2008 Aug 11. PMID 18695017